CLINICAL TRIAL: NCT02962388
Title: A Randomized, Multicenter Phase IIb Study to Evaluate the Efficacy and Safety of Ruxolitinib Versus Best Available Therapy in Patients With High Risk Essential Thrombocythemia, Who Are Resistant or Intolerant to Hydroxyurea: A FIM Study
Brief Title: The Ruxolitinib Versus Best Available Therapy Trial in Patients With High Risk ET in Second Line
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: not enough recruitment
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUXBETA trial
Record Dates: First submitted 2016-10-05; First posted 2016-11-11 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Essential Thrombocythemia
Keywords: efficacy; safety
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference therapy arm (Active Comparator): Best Available Therapy (BAT) in second line, after hydroxyurea. BAT restricted to anagrelide or IFNα/ PegIFNα in the study, according to the investigator decision
  Interventions: Drug: Anagrelide; Drug: IFNα/ PegIFNα
- Investigational therapy arm (Experimental): Ruxolitinib JAKAVI® Starting dose 10 mg BID, orally. To be increased or decreased (5 or 10 mg steps) per standardized dosing paradigm.
  Maximum dose 25 mg BID.
  Interventions: Drug: Ruxolitinib (JAKAVI®)

INTERVENTIONS:
Drug: Anagrelide — Anagrelide in the study, according to the investigator decision fom day 1 to 48 months
  Other Names: ARM A
  Arms: Reference therapy arm
Drug: Ruxolitinib (JAKAVI®) — Ruxolitinib (JAKAVI®) - Novartis. Tablets 5 mg. Starting dose 10 mg BID, orally. To be increased or decreased (5 or 10 mg steps) per standardized dosing Maximum dose 25 mg BID. fom day 1 to 48 months
  Other Names: ARM B
  Arms: Investigational therapy arm
Drug: IFNα/ PegIFNα — IFNα/ PegIFNα in the study, according to the investigator decision fom day 1 to 48 months
  Other Names: ARM A
  Arms: Reference therapy arm

SUMMARY:
Prospective national multicenter randomized open label phase IIb RUXBETA trial.

DETAILED DESCRIPTION:
A randomized, open label, multicenter phase IIb study to evaluate the efficacy and safety of Ruxolitinib versus best available therapy in patients with high risk essential thrombocythemia, who are resistant or intolerant to hydroxyurea.

ELIGIBILITY:
Inclusion Criteria:

Target Population

* Men and women, age more than or equal18 years and less than 75 years.
* Confirmed diagnosis of Essential Thrombocythemia for at least 6 months, according to the 2008 WHO criteria, with a high-risk status.
* Patients must have a treatment history for ET that meet the definition of resistance or intolerance to hydroxyurea therapy according to the ELN criteria as follow:

  * Platelets more than 600.0109/L after 3 months (12 weeks) of treatment at a dose over 2g/day.
  * Platelets more than 400.0 109/L and WBC less than 2.5109/L, whatever the dose of HU.
  * Platelets more than 400.0 109/L and Hb less than 10g/dl whatever the dose of HU.
  * Leg ulcers or other unacceptable muco-cutaneous toxicity.
  * HU-related fever.
* ECOG Performance Status (ECOG PS) less than or equal 2 at screening and at baseline.

Adequate Organ Function:

* Direct bilirubin less than 2.0 times the institutional Upper Limit of Normal (ULN).
* Hepatic enzymes (AST, ALT) less than or equal 2.5 times the institutional ULN.
* Adequate renal function at screening as demonstrated by MDRD-eGFR more than 30 mL/min/1.73m2.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy during and after the study.

  * A male subject of fathering potential must use an adequate method of contraception to avoid conception during and after the study to minimize the risk of pregnancy.
  * For females and males, these restrictions apply for 24 hours after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin hCG pregnancy test at Screening.
* Signed Written Informed Consent.
* Health insurance coverage.

Exclusion Criteria:

* Patients with thrombocytosis related to another MPN than ET
* Patients previously treated with a JAK2 inhibitor, Anagrelide or Interferon-alpha and prior history of therapy other than Hydroxyurea
* Contraindication to Ruxolitinib, Anagrelide or Interferon-alpha (if no eligible for anagrelide), hypersensitivity to an excipient

Medical history and concurrent diseases:

* Clinically significant cardiac disease (NYHA Class III or IV).
* Chronic hepatocellular disease.
* Subjects with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Ruxolitinib
* Subjects with clinically significant bacterial, fungal, parasitic or viral infection which requires therapy:

  * Subjects with acute bacterial infections requiring antibiotic use should delay screening/enrolment until the course of antibiotic therapy has been completed.
  * Subjects with active hepatitis A, B or C or with HIV positivity at screening.
  * Subjects with diagnosed primary immunodeficiency syndromes such as X-Linked a gammaglobulinemia and common variable immune deficiency.
  * Subject with medical history of tuberculosis
* History of progressive multifocal leucoencephalopathy (PML).
* Other malignant disease during the last 5 years prior to the inclusion except treated cervical intraepithelial neoplasia, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin, with no evidence for recurrence in the past 3 years.
* History of significant bleeding disorder not related to the ET.

  * Diagnosed congenital bleeding disorders,
  * Diagnosed acquired bleeding disorder within one year (e.g. acquired anti-factor VIII antibodies),
  * Ongoing or recent (3 months) significant gastrointestinal bleeding.
* Subjects with an uncontrolled undercurrent illness or any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
* Subjects being treated concurrently with a potent systemic inhibitor of CYP3A4 at the time of screening.
* Subjects being treated concurrently with any prohibited medications.
* Women who are pregnant or breastfeeding are not eligible for this study.
* Inability to freely provide consent through judiciary or administrative condition.
* Ongoing participation to another clinical investigational study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Failure-free patients | month 12
  Failure is defined by the occurrence of either intolerance and/or resistance to the second line therapy according to the protocol criteria

SECONDARY OUTCOMES:
Complete hematologic response | 48 months
  Number of Participants With normal Laboratory Values
AE/SAE | 48 months
  Rates, types and grades of AE/SAE related to the therapy, according to the NCI-CTCAE v4.0 classification
Median dose | 48 months
  Median dose of the treatment received
Thrombotic and hemorrhagic events | 48 months
  Cumulative incidence of thrombotic and hemorrhagic events incidence of progression into PV, secondary MF and MDS/acute leukemia
Quality of life questionnaire | 48 months
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane GIRAUDIER, MD PD, Principal Investigator — France Intergroupe Syndromes Myéloprolifératifs; LYDIA ROY, MD, Principal Investigator — France Intergroupe Syndromes Myéloprolifératifs
Locations (1):
- FILO, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
e crf

REFERENCES:
- See also: FILO site — http://www.filo-leucemie.org